CLINICAL TRIAL: NCT00209066
Title: A Means to Enhanced Cardiovascular Outcomes: Reduction of Exaggerated Platelet Activity Through Treatment of Depression.
Brief Title: Treatment of Reduced Heart Rate Variability Associated With Major Depression With Electroconvulsive Therapy
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: The Dana Foundation (Other)
Responsible Party: Principal Investigator, Dominique Musselman, Associate Professor, Emory University
Other Study IDs: 0422-1998; 98052113 (Other: Other)
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Electroconvulsive Therapy; Platelet Activation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate alterations in sympathetic tone in patients with major depression with and without ischemic heart disease and then to reevaluate these patients after 8 treatments with electroconvulsive therapy(ECT). We expect to support the hypothesis that HRV are pathophysiologically associated with the state of major depression. We hypothesize the following:

1. Heart rate variability (HRV) will be decreased prior to treatment of depression in comparison to post-treatment measures of HRV.
2. After 8 treatments with ECT, HRV will be increased under basal conditions.

DETAILED DESCRIPTION:
There is considerable evidence that patients with ischemic heart disease (IHD) and concurrent major depression have a less favorable prognosis than patients with IHD alone. Indeed, a number of recent studies implicate major depression in the pathophysiologic progression of cardiovascular disease as an independent risk factor, rather than a reaction to cardiovascular illness. This conclusion is supported by multiple recent studies (Anda et al; 1993; Markowitz and Matthews, 1991; Musselman et al., 1994, 1995).

Increased sympathetic tone and subsequent diminished heart rate variability secondary to elevated circulating levels of catecholamines provides a possible pathophysiologic link between IHD and depression. For example, Carney et al (1988) have established the correlation of increased heart rate and decreased heart rate variability (HRV) in patients with major depression and IHD. Thus it follows that enhancement of sympathetic tone may be important in the independent development of IHD and major depression. The interplay among these systems remains to be investigated. The present study seeks to determine the relationship between major depression and sympathetic tone.

The primary objective of the Research Protocol is to determine the effects of major depressive disorder (MDD) (see Specific Aim 1), and its treatment, on autonomic function (see Specific Aim 2). Twenty-five depressed patients with and 25 depressed patients without a history of ischemic cardiovascular disease will be recruited to this study.

To be determined is whether the exaggerated platelet reactivity and diminished HRV exhibited by depressed patients are affected by treatment with ECT. Autonomic function in depressed patients will be studied longitudinally before and after ECT. Heart rate variability (HRV) in depressed patients who exhibit a therapeutic response to ECT and who exhibited diminished HRV prior to treatment will support the hypothesis that HRV are pathophysiologically associated with the state of major depression. Successful ECT treatment of depressed mood that is not associated with normalization of HRV may indicate that: a) HRV is unrelated to Major Depressive Disorder, or b) HRV may reflect a pre-existing "trait" phenomena of major depressive disorder, or c) directly improve HRV.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Patients will not be accepted into the study if they abuse alcohol or drugs.

Patients will be excluded from the study if they have had an MI within the past three months, unstable crescendo angina or ongoing warfarin treatment

Patients also will not be accepted into the study if ECT will be harmful to them. These patients include:

1. those who have had a recent MI (<3 months)
2. those who have an infection of the brain,
3. those who have a condition in which there is increased intracranial pressure (e.g. a brain tumor)
4. those who cannot tolerate general anesthesia.

Any patient with a current DSM-IV Axis I diagnosis other than major depression will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with major depressive disorder presenting for a course of electroconvulsive therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 1998-11; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Dominique L Musselman, MD,MS, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Result] Royster EB, Trimble LM, Cotsonis G, Schmotzer B, Manatunga A, Rushing NN, Pagnoni G, Auyeung SF, Brown AR, Schoenbeck J, Murthy S, McDonald WM, Musselman DL. Changes in heart rate variability of depressed patients after electroconvulsive therapy. Cardiovasc Psychiatry Neurol. 2012;2012:794043. doi: 10.1155/2012/794043. Epub 2012 Aug 27. PMID 22966422